CLINICAL TRIAL: NCT01937845
Title: Evaluating the Health Outcomes of the Joslin Why WAIT? Program (Weight Achievement & Intensive Treatment Program)
Brief Title: Evaluating the Health Outcomes of the Joslin Why WAIT? Program
Status: Active, not recruiting | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Other Study IDs: CHS#: 06-26
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Evaluating the health outcomes of patients that were enrolled in Joslin's Why WAIT Program. These outcomes include BMI, A1C, lipid profile.

DETAILED DESCRIPTION:
This study is aimed to evaluate the health outcomes of patients enrolled in Joslin's Why WAIT Program. This program aims to control diabetes and help patients lose weight.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes with BMI over 35

Exclusion Criteria:

* Patients with type 1 diabetes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 diabetes enrolled in the Why WAIT? Program
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2006-08; Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Weight loss of 7% body weight | 13 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamdy O, Mottalib A, Morsi A, El-Sayed N, Goebel-Fabbri A, Arathuzik G, Shahar J, Kirpitch A, Zrebiec J. Long-term effect of intensive lifestyle intervention on cardiovascular risk factors in patients with diabetes in real-world clinical practice: a 5-year longitudinal study. BMJ Open Diabetes Res Care. 2017 Jan 4;5(1):e000259. doi: 10.1136/bmjdrc-2016-000259. eCollection 2017. PMID 28090332